CLINICAL TRIAL: NCT00707759
Title: Multicenter, Open-Label, Randomized Study on Steroid-Free Immunosuppression, in Comparison With Daily Steroid Therapy, in Pediatric Renal Transplant : Impact on Growth, Bone Metabolism and Acute Rejection
Brief Title: Steroid Withdrawal in Pediatric Renal Transplant: Impact on Growth, Bone Metabolism and Acute Rejection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Principal Investigator, Maria Angela Delucchi Bicocchi, Physician, Fondo Nacional de Desarrollo Científico y Tecnológico, Chile
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fondecyt1080166
Record Dates: First submitted 2008-06-26; First posted 2008-07-01 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-10

CONDITIONS: Kidney Diseases
Keywords: Pediatric renal transplantation,Bone metabolism (DXA-pQCT); mRNAFOXP3/IL-17,Steroid withdrawal
MeSH Terms: conditions — Kidney Diseases | interventions — Tacrolimus; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: withdrawal steroids (Experimental): Arms A: TAC + MMF + withdrawal steroids over a six-days following randomization.
  1°day: Methylprednisolone iv, 2-3 mg/kg/d 3 doses
  2ºday: Methylprednisolone iv, 2-3 mg/kg/d 3 doses
  3°day: Prednisone 2 mg/kg/d in 2 doses
  4ºday: Prednisone 1 mg/kg/d in 2 doses
  5ºday: Prednisone 0.5 mg/kg/d in 2 doses
  6ºday: Prednisone 0.25 mg/kg/d in 2 doses
  7ºday: Stop Prednisone
  Interventions: Drug: Tacrolimus (TAC)+ Mycophenolate Mofetil (MMF) + Withdrawal Prednisone
- B (Active Comparator): Arms B: TAC + MMF + prednisolone (see schedule)/day
  10°days after Tx: 2 mg/kg/d
  Day 11 - 20: 1 mg/kg/d
  Day 21 - 30: 0.5 mg/kg/d
  Day 31 - 60: 0.3 mg/k/d
  Week 8 - 12: 0.25 mg/k/d
  Week 12 - 16: 0.20 mg/k/d
  Week 16 - 20: 0.15 mg/k/d
  Month 6 - 12: 0.10 - 0.12 mg/k/d
  Interventions: Drug: Tacrolimus (TAC)+ Mycophenolate Mofetil (MMF) + prednisolone

INTERVENTIONS:
Drug: Tacrolimus (TAC)+ Mycophenolate Mofetil (MMF) + Withdrawal Prednisone — Arms A: Tacrolimus (TAC)+ Mycophenolate Mofetil (MMF) + withdrawal steroids over a six-days following randomization.
  1°day: Methylprednisolone iv, 2-3 mg/kg/d 3 doses
  2ºday: Methylprednisolone iv, 2-3 mg/kg/d 3 doses
  3°day: Prednisone 2 mg/kg/d in 2 doses
  4ºday: Prednisone 1 mg/kg/d in 2 doses
  5ºday: Prednisone 0.5 mg/kg/d in 2 doses
  6ºday: Prednisone 0.25 mg/kg/d in 2 doses
  7ºday: Stop Prednisone
  Arms: A: withdrawal steroids
Drug: Tacrolimus (TAC)+ Mycophenolate Mofetil (MMF) + prednisolone — Arms B: Tacrolimus (TAC)+ Mycophenolate Mofetil (MMF) + prednisolone (see schedule)/day
  10°days after Tx: 2 mg/kg/d
  Day 11 - 20: 1 mg/kg/d
  Day 21 - 30: 0.5 mg/kg/d
  Day 31 - 60: 0.3 mg/k/d
  Week 8 - 12: 0.25 mg/k/d
  Week 12 - 16: 0.20 mg/k/d
  Week 16 - 20: 0.15 mg/k/d
  Month 6 - 12: 0.10 - 0.12 mg/k/d
  Arms: B

SUMMARY:
The present study investigates the safety and efficacy of steroid withdrawal at six days post-transplant in pediatric renal recipients under concomitant immunosuppression based on antibodies anti IL2 (interleukin 2), Tacrolimus (TAC) and Mycophenolate Mofetil (MMF). To investigate the impact of this protocol in growth, bone metabolism, insulin- sensitivity and evaluate the expression of IL17 (interleukin 17) and mRNA FOXP3 (messenger ribonucleic acid forkhead box protein 3) as early markers of acute rejection (blood, urine and renal biopsy).

Hypothesis:Steroid withdrawal in renal pediatric transplant patients improves growth and bone metabolism without increasing the risk of acute rejection. The expression of FoxP3/IL17 in urine cells could be an early molecular markers of acute rejection.

DETAILED DESCRIPTION:
The intention of this investigation is to evaluate a prospective immunosuppressive protocol based on antibodies anti IL-2 (Ac-IL-2), Tacrolimus (TAC) and Mycophenolate Mofetil (MMF)and withdrawal steroids in renal transplant and to compare with a steroid-based protocol.

Objectives:

1. To evaluate growth and the impairment in the GH/IGF (growth hormone/insulin like growth factor) axis
2. To determine the impact of steroids on bone metabolism (biochemical parameters, DXA and pQCT)
3. To determine the steroid effect on metabolic factors (dyslipidemia, insulin- sensitivity and arterial hypertension)
4. To determine acute rejection incidence (protocol renal biopsy)
5. To evaluate the expression of IL-17 and mRNA FoxP3 as early markers of acute rejection (blood, urine and renal biopsy).

Two treatment regimes (Arms)will be compared in randomized form in the course of 12 months after transplantation.

Arm A: TAC + MMF + withdrawal of steroids over a six-days following randomization.

Arm B: TAC + MMF + prednisolone (see schedule)/day

ELIGIBILITY:
Inclusion Criteria:

* Age < 16.0 years
* Bone age of boys < 15 years, of girls < 13 years
* Prepuberal Tanner Status I
* First or second kidney transplant, living or deceased kidney donation
* Immunosuppression with Tacrolimus (TAC),Mycophenolate mofetil (MMF)
* Patients and parents, respectively, have given their written consent after enlightenment (informed consent)

Exclusion Criteria:

* Irreversible rejection of former transplant
* Highly reactive (> 30%) lymphocytotoxic antibodies within 12 months prior to transplantation
* Suspected insufficient medication compliance in dialysis
* Patients receiving a basic immunosuppression other than that prescribed in this protocol
* Simultaneous therapy with growth hormone after renal transplant

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2008-06; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Angela Delucchi, MD, Principal Investigator — Calvo Mackenna Children´s Hospital-University of Chile
Locations (1):
- Calvo Mackenna Children Hospital, Santiago, Metropolitan Region, Chile

RESULTS

PARTICIPANT FLOW:
Groups:
- A: Withdrawal Steroids: Arms A: TAC + MMF + withdrawal steroids over a six-days following randomization.
  1°day: Methylprednisolone iv, 2-3 mg/kg/d 3 doses
  2ºday: Methylprednisolone iv, 2-3 mg/kg/d 3 doses
  3°day: Prednisone 2 mg/kg/d in 2 doses
  4ºday: Prednisone 1 mg/kg/d in 2 doses
  5ºday: Prednisone 0.5 mg/kg/d in 2 doses
  6ºday: Prednisone 0.25 mg/kg/d in 2 doses
  7ºday: Stop Prednisone
  Tacrolimus (TAC)+ Mycophenolate Mofetil (MMF) + Withdrawal Prednisone: Arms A: Tacrolimus (TAC)+ Mycophenolate Mofetil (MMF) + withdrawal steroids over a six-days following randomization.
  1°day: Methylprednisolone iv, 2-3 mg/kg/d 3 doses
  2ºday: Methylprednisolone iv, 2-3 mg/kg/d 3 doses
  3°day: Prednisone 2 mg/kg/d in 2 doses
  4ºday: Prednisone 1 mg/kg/d in 2 doses
  5ºday: Prednisone 0.5 mg/kg/d in 2 doses
  6ºday: Prednisone 0.25 mg/kg/d in 2 doses
  7ºday: Stop Prednisone
- B: Control Steroids: Arms B: TAC + MMF + prednisolone (see schedule)/day
  10°days after Tx: 2 mg/kg/d
  Day 11 - 20: 1 mg/kg/d
  Day 21 - 30: 0.5 mg/kg/d
  Day 31 - 60: 0.3 mg/k/d
  Week 8 - 12: 0.25 mg/k/d
  Week 12 - 16: 0.20 mg/k/d
  Week 16 - 20: 0.15 mg/k/d
  Month 6 - 12: 0.10 - 0.12 mg/k/d
  Tacrolimus (TAC)+ Mycophenolate Mofetil (MMF) + prednisolone: Arms B: Tacrolimus (TAC)+ Mycophenolate Mofetil (MMF) + prednisolone (see schedule)/day
  10°days after Tx: 2 mg/kg/d
  Day 11 - 20: 1 mg/kg/d
  Day 21 - 30: 0.5 mg/kg/d
  Day 31 - 60: 0.3 mg/k/d
  Week 8 - 12: 0.25 mg/k/d
  Week 12 - 16: 0.20 mg/k/d
  Week 16 - 20: 0.15 mg/k/d
  Month 6 - 12: 0.10 - 0.12 mg/k/d
Period: Overall Study
Arm/Group | A: Withdrawal Steroids | B: Control Steroids
Started | 14 | 14
Completed | 12 | 12
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Withdrawal Steroids | B: Control Steroids | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.0 (3.3) | 6.9 (3.9) | 6.5 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  Chile | 12 | 12 | 24
Height Z-score [Mean (Standard Deviation); unit: units on a scale] | -2.5 (1.0) | -2.0 (1.2) | -2.3 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Stimulation of Growth After 12 Months (Delta Z-score)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A: Withdrawal Steroids | B: Control Steroids
Number analyzed (Participants) | 12 | 12
units on a scale | 1.2 (0.2) | 0.6 (0.1)

2. Secondary Outcome: Growth-factors (IGF-I, IGFBP-3) Bone Metabolism (FA, Ca/Cru, CaxP, 25(OH)VitD, FGF23, Klotho, PTH, DXA, pQCT) Insulin-sensitivity by ISI Method. Molecular Markers - Acute Rejection (FOXP3/IL-17). Acute Rejection Incidence/Protocol Renal Biopsy
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | A: Withdrawal Steroids | B: Control Steroids
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes